CLINICAL TRIAL: NCT07139457
Title: Wearable Epileptic Seizure Prediction and Alert Glasses Based on Neuromorphic Computing
Acronym: WESPG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MoH/CSR/25/29835; Khoula Hospital (Other: Oman MoH)
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy; Epileptic Seizures; Focal Epilepsy
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsies, Partial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (3):
- Young adults (Experimental): Participants aged 18-30 (equal male and female distribution) who will wear the NEXA seizure prediction glasses during both hospital-monitored and daily-life phases. Intervention involves continuous EEG monitoring, real-time seizure prediction, and alert notifications.
  Interventions: Device: Wearable seizure prediction and alert glasses
- middle-aged adults (Experimental): Participants aged 31-60 (equal male and female distribution) who will wear the NEXA seizure prediction glasses during both hospital-monitored and daily-life phases. Intervention involves continuous EEG monitoring, real-time seizure prediction, and alert notifications.
  Interventions: Device: Wearable seizure prediction and alert glasses
- Elderly adults (Experimental): Participants aged 60+ (equal male and female distribution) who will wear the NEXA seizure prediction glasses during both hospital-monitored and daily-life phases. Intervention involves continuous EEG monitoring, real-time seizure prediction, and alert notifications.
  Interventions: Device: Wearable seizure prediction and alert glasses

INTERVENTIONS:
Device: Wearable seizure prediction and alert glasses — A glasses-based wearable EEG system using the international 10-20 electrode placement standard with 4 dry spiked electrodes at F7, F8, T3 and T4. The device integrates neuromorphic computing for real-time seizure prediction, an artifact removal algorithm, and multi-modal alerts (vibration, light, sound). Data is logged for model improvement. The system is intended for continuous use in both hospital-monitored and daily-life settings.
  Other Names: NEXA glasses; wearable EEG glasses; neuromorphic seizure prediction device

SUMMARY:
The NEXA study aims to evaluate a new wearable EEG device designed as smart glasses with dry electrodes positioned according to the 10-20 system. The device captures real-time brain signals to detect patterns that may predict seizures, helping people with epilepsy. This study will test the device's safety, performance, and usability before seeking regulatory approval, including FDA clearance. The NEXA device is investigational and not yet approved by the U.S. FDA. The study will involve human participants who will wear the device while data is collected and analyzed. Results will help improve the device and support future certification for medical use.

DETAILED DESCRIPTION:
The NEXA Study is a prospective observational clinical trial designed to evaluate the safety, comfort, and performance of the NEXA wearable EEG device in patients with epilepsy. NEXA uses an innovative dry electrode system (two dome-shaped electrodes at the front and two spiked electrodes above the ears) aligned with the 10-20 EEG placement system to capture high-quality brain signals without the need for gels. The device integrates real-time artifact removal algorithms and a low-power neuromorphic chip for seizure detection and prediction. The study will compare NEXA's performance against standard EEG monitoring in hospital settings across Oman, with the primary goal of determining its accuracy in seizure detection and prediction. Secondary outcomes include electrode comfort, usability, compliance, and safety. Data from this study will support regulatory submissions and demonstrate NEXA's potential as a practical and reliable solution for continuous EEG monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with a confirmed epilepsy diagnosis by a neurologist or epilepsy specialist.
* History of active seizures within the last year, under stable treatment (medications, VNS, diet, or surgery) for at least 3 months.
* Capacity to provide informed consent (or via legal representative if cognitively impaired).
* Willingness to participate and sign consent.
* Residents of Oman attending Khoula Hospital or affiliated clinics.
* Stable general health without acute or severe comorbidities.
* Ability and willingness to attend study visits and follow protocols.

Exclusion Criteria:

* Seizures from non-epileptic causes (e.g., psychogenic, metabolic, tumors).
* Under 18 years of age.
* Severe cognitive impairment preventing consent or protocol adherence.
* Pregnant or planning pregnancy during the study.
* Severe uncontrolled medical conditions (e.g., heart disease, cancer).
* History of non-compliance with epilepsy treatment or follow-ups.
* Severe psychiatric disorders affecting participation or safety.
* History of substance abuse interfering with study adherence.
* Known allergies or hypersensitivity to study medications or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accurate Seizure Detection in Real-World Patient Settings | From start of patient data collection until end of clinical trial (estimated 3 months).
  Measure the ability of the NEXA wearable EEG glasses to detect epileptic seizures in real-world patient settings with a target accuracy of ≥95%, using simultaneous hospital EEG recordings as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Said Al-Mawali, PhD, Principal Investigator — Oman Ministry of Health
Locations (1):
- Khoula Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: No
Sharing is on permission basis based on Omani Ministry of Health policies.